CLINICAL TRIAL: NCT04709627
Title: Verification of Clinical Utility: enFlow IV Fluid and Blood Warming System
Brief Title: enFlow IV Fluid and Blood Warming System
Status: Completed | Type: Observational
Sponsor: Vyaire Medical (Industry)
Collaborators: Helsinki University Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 100-P0093; 30000000064) (Other: Vyaire Medical)
Record Dates: First submitted 2021-01-08; First posted 2021-01-14 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Hypothermia; Anesthesia
Keywords: Surgery
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- 60 minute surgery: Patients completing at least 60 minutes of surgery
  Interventions: Device: enFlow IV Fluid and Blood Warming System

INTERVENTIONS:
Device: enFlow IV Fluid and Blood Warming System — The enFlow IV fluid/blood warming system's intended use is for warming blood, blood products and intravenous solutions prior to administration.

SUMMARY:
This study is part of a post-market clinical follow-up (PMCF). The purpose of this study is to verify in a routine clinical environment with a number of caregivers and subjects that the enFlow performs as intended when used as an element of maintaining acceptable core temperatures.

DETAILED DESCRIPTION:
Eligible subjects from the study will be recruited from patients with scheduled surgeries. After being informed about the study and potential risks, patients given informed consent will undergo scheduled surgery with the use of enFlow IV Fluid and Blood Warming System. The following temperature measurements will be collected during surgery:

* Baseline temperature measurement (0-15 minutes prior to induction)
* Induction temperature measurements (15 minutes, 30 minutes, 60 minutes, 90 minute post-induction)
* Continued temperature measurements (every 30 minutes, plus end of surgery)
* OR ambient temperature at induction and end of surgery.

Temperature will be measured and collected post-surgery upon arrival to the PACU and 30 minutes post-arrival.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients requiring surgery expected to last at least 1 hour.
* Expectation of the perioperative need for at least one liter of infused fluids warmed during infusion
* Informed Consent

Exclusion Criteria:

* Recent history of fever (>38 C, within 24 hours of surgery)
* Active infection
* Pregnant women
* Terminal illness (<30 days)
* Intended use of cardiopulmonary bypass
* Clinical intention for perioperative cooling and hypothermia
* unavailability of esophageal measurement during surgery
* Attending physician does not believe participation of the patient is in their best interest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects from the study will be recruited from patients with scheduled surgeries. Most are expected to be inpatient due to the exclusion of short surgeries. For this study, only adults will be enrolled. Participation will also be limited to patients fluent in the language(s) of the information and consent form.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Maintenance of intraoperative core temperature | 15 and 30 minutes post-induction, then every 30 minutes untl the termination of the scheduled surgical procedure, and a final measurement recorded at the time of termination of the scheduled surgical procedure.
  Core temperature is defined as the highest temperature reading during 30 seconds made within 5 minutes of protocol time. The primary outcome measure will be the mean of the temperature measurements taken during the course of surgery

SECONDARY OUTCOMES:
Core temperature for two periods | Induction: first 90 minutes. Post-Induction: after 90 minutes until the end of surgery,
  The mean of the measurements taken during the Induction period and during the Post-Induction period.
Number of hypothermic events | During 30 seconds made within 5 minutes of protocol time
  The incidence and duration of hypothermic events (<36.0C).
Number of hyperthermic events | During 30 seconds made within 5 minutes of protocol time
  The incidence and duration of hyperthermic events (>38.0 oC).
Incidence of infusate outside acceptable operating range (i.e., device "green range") | Induction: first 90 minutes. Post-Induction: after 90 minutes until the end of surgery,
  Device reading 35-42 oC

CONTACTS AND LOCATIONS:
Overall Officials: Mikko Lax, MD, Principal Investigator — Helsinki and Uusimaa Hospital District, Helsinki University Hospital; Seppo Mustola, MD, PhD, Principal Investigator — South Karelia Central Hospital (EKSOTE, ALTEK), Dept. of Anesthesiology
Locations (2):
- Finland (2):
  - Helsinki and Uusimaa Hospital District, Helsinki University Hospital, Helsinki
  - South Karelia Central Hospital (EKSOTE, ALTEK), Lappeenranta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Campbell G, Alderson P, Smith AF, Warttig S. Warming of intravenous and irrigation fluids for preventing inadvertent perioperative hypothermia. Cochrane Database Syst Rev. 2015 Apr 13;2015(4):CD009891. doi: 10.1002/14651858.CD009891.pub2. PMID 25866139
- [Background] National Institute of Health and Care Excellence (NICE). Hypothermia: prevention and management in adults having surgery Clinical guideline. Original Published: 23 April 2008. nice.org.uk/guidance/cg65 2019
- [Background] Pesonen E, Silvasti-Lundell M, Niemi TT, Kivisaari R, Hernesniemi J, Makinen MT. The focus of temperature monitoring with zero-heat-flux technology (3M Bair-Hugger): a clinical study with patients undergoing craniotomy. J Clin Monit Comput. 2019 Oct;33(5):917-923. doi: 10.1007/s10877-018-0227-z. Epub 2018 Nov 22. PMID 30467673
- [Background] Makinen MT, Pesonen A, Jousela I, Paivarinta J, Poikajarvi S, Alback A, Salminen US, Pesonen E. Novel Zero-Heat-Flux Deep Body Temperature Measurement in Lower Extremity Vascular and Cardiac Surgery. J Cardiothorac Vasc Anesth. 2016 Aug;30(4):973-8. doi: 10.1053/j.jvca.2016.03.141. Epub 2016 Mar 22. PMID 27521967